CLINICAL TRIAL: NCT00194519
Title: Phase III Randomized Placebo-Controlled Trial of HSV-2 Suppression to Prevent HIV Transmission Among HIV-Discordant Couples
Brief Title: Herpes Simplex Virus Type 2 (HSV-2) Suppression to Prevent HIV Transmission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Connie Celum, Prof of Medicine & Global Health, Adjunct Prof of Epidemiology, School of Medicine: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00000867; Gates Foundation Grant #26469; NCT00197574 (obsolete NCT alias); NCT00197600 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: HIV Infection; Herpes Simplex, Genital; Sexually Transmitted Diseases
Keywords: HIV infection; HIV transmission; genital herpes; sexual intercourse; sexual transmitted infection; acyclovir; HIV Seronegativity; Treatment Naive; HIV-discordant couples; HIV serodiagnosis
MeSH Terms: conditions — HIV Infections; Herpes Genitalis; Sexually Transmitted Diseases; Coitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acyclovir (Active Comparator)
  Interventions: Drug: Generic acyclovir
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Generic acyclovir — 400 mg twice-daily oral
  Arms: Acyclovir
Drug: Placebo — twice-daily oral
  Arms: Placebo

SUMMARY:
The University of Washington has received funding to conduct a proof-of-concept trial to assess the impact of suppression of genital herpes on HIV infectiousness. This study (the Partners in Prevention Study) will enroll HIV discordant heterosexual couples in which the HIV-infected partner is co-infected with herpes simplex virus type 2 (HSV-2) to test the efficacy of twice daily (bid) acyclovir (400 mg) given to the HIV-infected partner to prevent transmission to his/her HIV negative partner(s). This randomized, double-blind, placebo-controlled proof-of-concept trial will provide evidence for the efficacy of HSV-2 suppression with daily acyclovir on HIV transmission among HIV-discordant couples among whom the HIV-positive partner is also HSV-2 seropositive with CD4 >250. The researchers hypothesis is that, by decreasing the frequency and amount of genital HIV shedding, standard doses of daily acyclovir 400 mg bid will reduce the rate of HIV transmission by 50% in HIV-discordant couples among whom the HIV-infected partner is HSV-2 positive.

Under the study protocol version 4.1.1, 3000 HIV-discordant heterosexual couples in which the HIV-positive partner is HSV-2 positive and has a CD4 count >250 will be recruited; participants will be followed for up to 2 years. A 4% per year HIV incidence in the placebo arm is assumed.

The first study site began enrolling participants on 17 November 2005. As of September 2006, 14 sites in Eastern and Southern Africa had participated in recruiting the 2300 HIV-discordant couples enrolled to date.

DETAILED DESCRIPTION:
Herpes simplex virus type-2 (HSV-2) is the primary cause of genital ulcers and one of the most prevalent sexually transmitted diseases worldwide. Consistently, over 30 studies have found HSV-2 infection to be a risk factor for HIV acquisition with an overall relative risk of 2.1 in the studies that demonstrated HSV-2 preceded HIV infection. A recent study of HIV-discordant couples from Rakai, Uganda, has shown that at all levels of HIV viral load in the HIV-positive partner, HSV-2 infection in the susceptible partner increased the per-contact risk of acquisition of HIV five-fold, and GUD in the HIV-source partner increased the per-contact risk of HIV transmission five-fold. As strong as these epidemiological data are, an intervention trial is required to define the clinical and public health significance of these findings.

This trial will directly answer the extent to which HSV-2 infection increases infectiousness of HIV/HSV-2 co-infected persons and the relative reduction in HIV transmission among HSV-2 seropositive persons treated with daily suppressive antiviral therapy. Acyclovir has an acceptable safety profile for widespread STD treatment and is inexpensive, well-tolerated, and episodic and long-term suppressive therapy has not been associated with increased acyclovir resistance. Given high HSV-2 seroprevalence in HIV-infected persons (70-80%) and high HIV incidence in populations with high prevalence of HSV-2 infection worldwide, this approach could have great public health importance by providing a safe, acceptable, and cost-effective method to reduce HIV transmission among HIV-infected persons who are also HSV-2 seropositive.

Sites that have enrolled couples in this study include: Johannesburg (2 sites) and Cape Town, South Africa; Gaborone, Botswana; Kitwe/Ndola and Lusaka, Zambia; Nairobi, Kisumu, Eldoret and Thika, Kenya; Moshi, Tanzania; Kampala, Uganda; and Kigali, Rwanda.

ELIGIBILITY:
Inclusion Criteria:

Potential index (HIV-infected) participants must meet the following criteria (by self-report, unless otherwise indicated) in order to be eligible for inclusion in the study:

* Of legal age to provide independent informed consent for research per local regulations and guidelines.
* Able and willing to provide written informed consent to be screened for and to take part in the study. (Note: Index participants who are not willing to provide genital tract specimens for HIV viral load quantitation, but are willing to undergo all other study procedures, will be considered eligible for inclusion in the study.)
* Part of a heterosexual couple in which one partner meets the study eligibility criteria for index participants and the other partner meets the study eligibility criteria for partner participants. Couples are defined as partners who are sexually active and plan to remain in the relationship for at least one year. Each site will develop appropriate criteria for determining whether a couple is likely to remain in the relationship (i.e., married, duration of partnership, cohabitation, have children).
* Has had vaginal intercourse with the partner participant at least three times in the last three months.
* Plans to maintain his/her relationship with the partner participant for the next 24 months.
* HIV-infected based on positive EIA.
* HSV-2-seropositive based on the Focus HSV-2 EIA (performed by study staff) with an index ratio of at least 3.5 or if Focus EIA IN 1.1-3.4, confirmed by HSV-2 WB dot-blot performed at the UW.
* CD4 cell count (performed by study staff) of at least 250 cells/mm3.
* No history of any clinical AIDS-defining diagnoses.
* Able and willing to provide adequate locator information for study retention purposes, as defined by local standard operating procedures.

Potential partner (HIV-uninfected at enrollment) participants must meet the following criteria (by self-report, unless otherwise indicated) in order to be eligible for inclusion in the study:

* Of legal age to provide independent informed consent for research per local regulations and guidelines.
* Able and willing to provide written informed consent to be screened for and to take part in the study.
* Part of a heterosexual couple in which one partner meets the study eligibility criteria for index participants and the other partner meets the study eligibility criteria for partner participants.
* Has had vaginal intercourse with the study partner at least three times in the last three months.
* Plans to maintain his/her relationship with the index participant for the next 24 months.
* HIV-uninfected based on negative HIV EIA tests.
* Able and willing to provide adequate locator information for study retention purposes, as defined by local standard operating procedures.

Exclusion Criteria:

Potential index (HIV-infected) participants who meet any of the following criteria (by self-report, unless otherwise indicated) will be excluded from the study:

* Current use of combination antiretroviral therapy
* Known history of adverse reaction to acyclovir.
* Known history of persistent genital ulcers unresponsive to episodic acyclovir therapy.
* Known plans to re-locate or travel away from the study site for more than two consecutive months during the next 24 months.
* Pregnant, based on participant self-report or urine testing performed by study staff. (Note: Self-reported pregnancy is adequate for exclusion from the study. A documented negative test performed by study staff is required for inclusion.)

Potential partner participants who meet any of the following criteria (by self-report, unless otherwise indicated) will be excluded from the study:

* Has had sexual intercourse with a partner other than the index participant in the last two months.
* Known plans to re-locate or travel away from the study site for more than two consecutive months during the next 24 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3408 (Actual)
Dates: Start 2004-11; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Sequence-verified HIV-transmission from index to partner participant | March 2009

SECONDARY OUTCOMES:
Measure effect of viral load, gender and other factors on HIV transmission | March 2009
Assess adherence to acyclovir suppressive therapy | March 2009
Assess effect of twice daily acyclovir on the frequency of genital ulcers | March 2009
Assess effect of twice daily acyclovir on plasma HIV viral load | March 2009
Assess effects of twice daily acyclovir on the sexual behaviors | March 2009
Assess host immunologic and virologic determinants of HIV transmission | March 2009

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD, MPH, Principal Investigator — University of Washington; Jairam Lingappa, MD, PhD,, Study Director — University of Washington; Anna Wald, MD, MPH, Study Chair — University of Washington
Locations (13):
- Botswana-Harvard Partnership, Gabarone, Botswana
- Kenya (4):
  - Moi University - Indiana University, Eldoret
  - Kemri - Ucsf, Kisumu
  - University of Nairobi, Nairobi
  - Partners Study Thika Site, Thika
- Projet San Francisco-Emory University, Kigali, Rwanda
- South Africa (3):
  - University of Cape Town, Cape Town
  - Perinatal HIV Research Unit, University of Witswatersrand, Johannesburg
  - Reproductive Health and HIV Research Unit, Johannesburg
- Kilimanjaro Christian Medical College-Harvard University, Moshi, Tanzania
- Mulago Hospital - IDI, Kampala, Uganda
- Zambia (2):
  - Zambia-Emory HIV Research Project, Lusaka
  - Zambia-Emory HIV Research Project, Ndola/Kitwe

REFERENCES:
- [Derived] Mackelprang RD, Bamshad MJ, Chong JX, Hou X, Buckingham KJ, Shively K, deBruyn G, Mugo NR, Mullins JI, McElrath MJ, Baeten JM, Celum C, Emond MJ, Lingappa JR; Partners in Prevention HSV/HIV Transmission Study and the Partners PrEP Study Teams. Whole genome sequencing of extreme phenotypes identifies variants in CD101 and UBE2V1 associated with increased risk of sexually acquired HIV-1. PLoS Pathog. 2017 Nov 6;13(11):e1006703. doi: 10.1371/journal.ppat.1006703. eCollection 2017 Nov. PMID 29108000
- [Derived] de Bruyn G, Magaret A, Baeten JM, Lingappa JR, Ndase P, Celum C, Wald A; Partners in Prevention HSV/HIV Transmission Study Team. Mortality in members of HIV-1 serodiscordant couples in Africa and implications for antiretroviral therapy initiation: results of analyses from a multicenter randomized trial. BMC Infect Dis. 2012 Oct 30;12:277. doi: 10.1186/1471-2334-12-277. PMID 23130818
- [Derived] Lingappa JR, Thomas KK, Hughes JP, Baeten JM, Wald A, Farquhar C, de Bruyn G, Fife KH, Campbell MS, Kapiga S, Mullins JI, Celum C; Partners in Prevention HSV/HIV Transmission Study Team. Partner characteristics predicting HIV-1 set point in sexually acquired HIV-1 among African seroconverters. AIDS Res Hum Retroviruses. 2013 Jan;29(1):164-71. doi: 10.1089/AID.2012.0206. PMID 23061422
- [Derived] Cohen CR, Lingappa JR, Baeten JM, Ngayo MO, Spiegel CA, Hong T, Donnell D, Celum C, Kapiga S, Delany S, Bukusi EA. Bacterial vaginosis associated with increased risk of female-to-male HIV-1 transmission: a prospective cohort analysis among African couples. PLoS Med. 2012;9(6):e1001251. doi: 10.1371/journal.pmed.1001251. Epub 2012 Jun 26. PMID 22745608
- [Derived] Mujugira A, Magaret AS, Baeten JM, Celum C, Lingappa J. Risk Factors for HSV-2 Infection among Sexual Partners of HSV-2/HIV-1 Co-Infected Persons. BMC Res Notes. 2011 Mar 15;4:64. doi: 10.1186/1756-0500-4-64. PMID 21406077
- [Derived] Campbell MS, Mullins JI, Hughes JP, Celum C, Wong KG, Raugi DN, Sorensen S, Stoddard JN, Zhao H, Deng W, Kahle E, Panteleeff D, Baeten JM, McCutchan FE, Albert J, Leitner T, Wald A, Corey L, Lingappa JR; Partners in Prevention HSV/HIV Transmission Study Team. Viral linkage in HIV-1 seroconverters and their partners in an HIV-1 prevention clinical trial. PLoS One. 2011 Mar 2;6(3):e16986. doi: 10.1371/journal.pone.0016986. PMID 21399681
- [Derived] Lingappa JR, Baeten JM, Wald A, Hughes JP, Thomas KK, Mujugira A, Mugo N, Bukusi EA, Cohen CR, Katabira E, Ronald A, Kiarie J, Farquhar C, Stewart GJ, Makhema J, Essex M, Were E, Fife KH, de Bruyn G, Gray GE, McIntyre JA, Manongi R, Kapiga S, Coetzee D, Allen S, Inambao M, Kayitenkore K, Karita E, Kanweka W, Delany S, Rees H, Vwalika B, Magaret AS, Wang RS, Kidoguchi L, Barnes L, Ridzon R, Corey L, Celum C; Partners in Prevention HSV/HIV Transmission Study Team. Daily acyclovir for HIV-1 disease progression in people dually infected with HIV-1 and herpes simplex virus type 2: a randomised placebo-controlled trial. Lancet. 2010 Mar 6;375(9717):824-33. doi: 10.1016/S0140-6736(09)62038-9. Epub 2010 Feb 12. PMID 20153888
- [Derived] Celum C, Wald A, Lingappa JR, Magaret AS, Wang RS, Mugo N, Mujugira A, Baeten JM, Mullins JI, Hughes JP, Bukusi EA, Cohen CR, Katabira E, Ronald A, Kiarie J, Farquhar C, Stewart GJ, Makhema J, Essex M, Were E, Fife KH, de Bruyn G, Gray GE, McIntyre JA, Manongi R, Kapiga S, Coetzee D, Allen S, Inambao M, Kayitenkore K, Karita E, Kanweka W, Delany S, Rees H, Vwalika B, Stevens W, Campbell MS, Thomas KK, Coombs RW, Morrow R, Whittington WL, McElrath MJ, Barnes L, Ridzon R, Corey L; Partners in Prevention HSV/HIV Transmission Study Team. Acyclovir and transmission of HIV-1 from persons infected with HIV-1 and HSV-2. N Engl J Med. 2010 Feb 4;362(5):427-39. doi: 10.1056/NEJMoa0904849. Epub 2010 Jan 20. PMID 20089951
- [Derived] Baeten JM, Donnell D, Kapiga SH, Ronald A, John-Stewart G, Inambao M, Manongi R, Vwalika B, Celum C; Partners in Prevention HSV/HIV Transmission Study Team. Male circumcision and risk of male-to-female HIV-1 transmission: a multinational prospective study in African HIV-1-serodiscordant couples. AIDS. 2010 Mar 13;24(5):737-44. doi: 10.1097/QAD.0b013e32833616e0. PMID 20042848
- [Derived] Guthrie BL, Kiarie JN, Morrison S, John-Stewart GC, Kinuthia J, Whittington WL, Farquhar C. Sexually transmitted infections among HIV-1-discordant couples. PLoS One. 2009 Dec 14;4(12):e8276. doi: 10.1371/journal.pone.0008276. PMID 20011596
- [Derived] Lingappa JR, Kahle E, Mugo N, Mujugira A, Magaret A, Baeten J, Bukusi EA, Cohen CR, Katabira E, Ronald A, Kiarie J, Farquhar C, Stewart GJ, Makhema J, Essex M, Were E, Fife K, Debruyn G, Gray G, McIntyre J, Manongi R, Kapiga S, Coetzee D, Allen S, Inambao M, Kayitenkore K, Karita E, Kanweka W, Delany S, Rees H, Vwalika B, Coombs RW, Morrow R, Whittington W, Corey L, Wald A, Celum C; Partners HSV-2/HIV-1 Transmission Study Team. Characteristics of HIV-1 discordant couples enrolled in a trial of HSV-2 suppression to reduce HIV-1 transmission: the partners study. PLoS One. 2009;4(4):e5272. doi: 10.1371/journal.pone.0005272. Epub 2009 Apr 30. PMID 19404392